CLINICAL TRIAL: NCT03719755
Title: Comparison of Urinary Tract Infections Rates Using 50% Dextrose Plus Washout Versus Normal Saline as Cystoscopy Fluid: a Prospective Study
Brief Title: Urinary Tract Infections Rates Using 50% Dextrose Plus Washout Versus Normal Saline as Cystoscopy Fluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johnny Yi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-000176
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant masked to distention media
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50% dextrose (Active Comparator): Cystoscopic distention of 40 cc of 50% dextrose plus 300 cc of normal saline washout
  Interventions: Procedure: 50% dextrose
- Normal Saline (Placebo Comparator): Cystoscopic distention media of normal saline.
  Interventions: Procedure: Normal Saline

INTERVENTIONS:
Procedure: 50% dextrose — maximum injection of 40 cc of 50% dextrose plus 300 cc of normal saline washout versus normal saline after hysterectomy for benign indications.
  Arms: 50% dextrose
Procedure: Normal Saline — Cystoscopic distention media of normal saline
  Arms: Normal Saline

SUMMARY:
Our study will compare the rates of postoperative urinary tract infections (UTI) between patients who undergo cystoscopy using 50% dextrose injection plus bladder washout versus normal saline after hysterectomy for benign indications. Primary outcome will be rates of urinary tract infections at 6-9 days post-operatively. This will be defined as a urine culture yielding greater than 100,000 gram-negative colony-forming units per milliliter.

DETAILED DESCRIPTION:
This will be a prospective cohort study of the rate of UTIs after cystoscopic distention media of normal saline with maximum injection of 40 cc of 50% dextrose plus 300 cc of normal saline washout versus normal saline after hysterectomy for benign indications.

A pre-operative urine culture will be obtained via mid-stream clean catch prior to administration of routine pre-operative prophylactic antibiotics.

At 6-9 days post-operatively, a repeat urine culture will be obtained via mid-stream clean catch. Appropriate treatment will be administered if the urine culture is positive.Primary outcome will be rates of urinary tract infections at 6-9 days post-operatively. This will be defined as a urine culture yielding greater than 100,000 gram-negative colony-forming units per milliliter.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative scheduling CPT codes for hysterectomy

Exclusion Criteria:

* Discharged home with indwelling foley catheter
* Indwelling foley catheter > 24 hours
* Ureteral injury
* Chronic immunosuppression
* History of diabetes
* Recurrent UTIs (≥2 infections in six months or ≥3 infections in one year)
* Reported Chronic Kidney Disease
* Renal anomalies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — hysterectomy for all indications
Enrollment: 152 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
rates of urinary tract infections at 6-9 days post-operative | 6-9 days post-operative
  be rates of urinary tract infections at 6-9 days post-operatively. This will be defined as a urine culture yielding greater than 100,000 gram-negative colony-forming units per milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Yi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials